CLINICAL TRIAL: NCT04733963
Title: A Phase II, Randomized, Controlled Study to Assess the Efficacy and Safety of Fruquintinib Plus Capecitabine Versus Bevacizumab Plus Capecitabine as Maintenance Treatment Following First-line Chemotherapy for Metastatic Colorectal Cancer
Brief Title: Fruquintinib Plus Capecitabine Versus Bevacizumab Plus Capecitabine as Maintenance Therapy Following First-line Treatment for Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Ying Yuan, MD, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRUCA
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Fruquintinib maintenance
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Maintenance therapy with Fruquintinib Plus Capecitabine
  Interventions: Drug: Fruquintinib Plus Capecitabine
- Arm B (Active Comparator): Maintenance therapy with Bevacizumab Plus Capecitabine
  Interventions: Drug: Bevacizumab Plus Capecitabine

INTERVENTIONS:
Drug: Fruquintinib Plus Capecitabine — Maintenance therapy with fruquintinib at the dose determined in phase safety lead-in, orally once daily, on d1-21, given every 4 weeks (Q4W); plus capecitabine at the dose 850mg/m2, orally twice daily, d1-7, given every 2 weeks (Q2W); until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal
  Arms: Arm A
Drug: Bevacizumab Plus Capecitabine — Maintenance therapy with bevacizumab at the dose 5mg/kg q2w (Q2W); plus capecitabine at the dose 850mg/m2, orally twice daily, d1-7, given every 2 weeks (Q2W); until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal
  Arms: Arm B

SUMMARY:
This is an open-label, multicenter, randomized phase 2 study evaluating the efficacy and safety of fruquintinib plus capecitabine versus bevacizumab plus capecitabine as maintenance therapy following first-line treatment for metastatic colorectal cancer. Patients who have already achieved disease control (including CR/PR and SD), without discontinuation for toxicity, and are progression free after 4-6 months of standard first-line induction treatment will be assigned to 2 maintenance treatment groups by randomization in a 1:1 ratio to receive fruquintinib + capecitabine (Arm A) or bevacizumab + capecitabine (Arm B). The study contains a safety lead-in phase in which the safety and tolerability of fruquintinib + capecitabine will be assessed prior to the phase 2 portion of the study. All patients from Arm A and Arm B will be treated until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal (whichever occurs earlier).

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old (including 18 and 75) at the time of signing the informed consent;
2. Patients who have been histologically or cytologically confirmed adenocarcinoma of the colon or rectum (stage IV);
3. Patients who have achieved disease control (including CR/PR and SD) after 4-6 months of first-line standard chemotherapy (FOLFOX, FOLFIRI, XELOX ± targeted therapy) and are progression free at the start of maintenance therapy;
4. At least one measurable metastatic lesion(s) as defined by RECIST version 1.1;
5. ECOG performance status of 0-1;
6. Body weight ≥40Kg;
7. LVEF≥50%;
8. Life expectancy≥3 months;
9. Adequate organ and bone marrow functions:

   Neutrophils >1.5×109/L, platelets >100×109/L, and hemoglobin >9 g/dL; Total bilirubin <1.5×upper limit of normal (ULN); aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <2.5×ULN (<5×ULN in case of liver metastases); Creatinine clearance (calculated according to Cockcroft and Gault) ≥50 mL/min; Urinary protein / creatinine ratio < 1 (or urine analysis < 1 + or 24-hour urinary protein < 1g / 24 h);
10. Able to take oral medication;
11. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration;
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Any factors that influence the usage of oral administration;
3. Those who have been proved to be allergic to fruquintinib and / or its excipients;
4. Blood transfusion was performed within 1 week before randomization;
5. Non-controlled hypertension after monotherapy, that is, systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg;
6. Intercurrence with one of the following: coronary artery disease, arrhythmia and heart failure;
7. Clinically significant electrolyte abnormality;
8. Proteinuria ≥ 2+ (1.0g/24hr);
9. Previous treatment with VEGFR inhibition;
10. Evidence of CNS metastasis;
11. Severe intolerance to capecitabine or 5-FU;
12. Disability of serious uncontrolled intercurrence infection;
13. Uncontrolled hemorrhage in GI;
14. Have evidence or a history of bleeding tendency within two months of the enrollment;
15. Abdominal fistula or gastrointestinal perforation occurred within 6 months before the first treatment, unless repaired by surgery;
16. Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including stroke and transient ischemic attack) , etc.;
17. Within 6 months before the first recruitment occurs acute myocardial infarction, acute coronary syndrome or CABG;
18. Incomplete healing of skin trauma, surgical site, wound site or severe mucosal ulcer. Bone fracture or wounds that was not cured for a long time;
19. APTT and /or PT >1.5×ULN;
20. Clinically detectable secondary primary malignancies at the time of enrollment, or had other malignancies in the past 5 years (excluding fully treated basal cell carcinoma of the skin or carcinoma in situ of the cervix);
21. Patients who are not suitable for the study judged by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From Baseline to primary completion date, about 2 years
  Progression-free survival is determined from the date of treatment to PD or death from any cause

SECONDARY OUTCOMES:
Overall Survival | From Baseline to primary completion date, about 2 years
  Overall survival is determined from the date of treatment to death from any cause or the last follow-up date
Adverse Events and Serious Adverse Events | From Baseline to primary completion date, about 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.
QoL | From Baseline to primary completion date, about 24 months
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.

OTHER OUTCOMES:
Exploratory Endpoint | From Baseline to primary completion date, about 24 months
  Explore any correlation between clinical outcomes and baseline characteristics, and biomarkers associated with the antitumor activity of fruquintinib based on blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No